CLINICAL TRIAL: NCT00463502
Title: The Effect of Metformin Treatment on Thyroid Hormone Metabolism in Euthyroid Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Haydarpasa Numune State Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 07-013
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Last update posted 2007-04-20 (Estimated); Status verified 2007-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: The purpose of study was investigated the effect of; metformin on thyroid hormone metabolism in euthyroid patients; with type 2 DM. The results revealed significant decreases; in TSH and fT4
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Metformin

SUMMARY:
Aim: To investigate the effects of metformin treatment on thyroid hormone metabolism in euthyroid patients with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* The patients included in this study were the ones who were newly diagnosed with type 2 diabetes mellitus

Exclusion Criteria:

* Presence of thyroid disorders, positive thyroid autoantibodies and usage of medications affecting thyroid hormones such as amiodarone, lithium were accepted as exclusion criterions

Ages: 35 Years to 78 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ozdemir, Principal Investigator — Unaffiliation